CLINICAL TRIAL: NCT03780270
Title: Preventive Treatment Approach of Early Caries Lesions With Contemporary Methods of Remineralization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Dentistry Clinical Center of Kosovo (Other)
Responsible Party: Principal Investigator, Dafina Doberdoli, Principal Investigator, University Clinical Centre of Kosova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 500
Record Dates: First submitted 2018-12-06; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Tooth Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Fluoride Varnish (Fluor Protector S; Ivoclar, 7'700 ppm F-) application at Day 0 and Day180.
  => Group: Fluoride Varnish
  Interventions: Device: Fluoride Varnish
- Test1 (Experimental): Single application of Curodont Repair (P11-4) at Day 0 followed by a Fluoride Varnish (Fluor Protector S; Ivoclar, 7'700 ppm F-) application. Another fluoride Varnish application at Day180.
  => Group: Curodont Repair + Fluoride Varnish
  Interventions: Device: Fluoride Varnish; Device: Curodont Repair
- Test2 (Experimental): Single application of Curodont Repair (P11-4) at Day 0. Curodont Protect (tooth gel containing P11-4 matrix) is handed out and subjects are asked to apply it 2x weekly at home after regular teeth cleaning in the evening for the whole study period (Day 360).
  => Group: Curodont Repair + Curodont Protect
  Interventions: Device: Curodont Repair; Device: Curodont Protect

INTERVENTIONS:
Device: Fluoride Varnish — Fluor Protector S (Ivoclar, 7'700 ppm F-)
  Arms: Control; Test1
Device: Curodont Repair — P11-4 (monomeric peptide) - for professional use
  Arms: Test1; Test2
Device: Curodont Protect — Tooth gel (containing P11-4 assembled to a fibrillary matrix) - for home use (OTC)
  Arms: Test2

SUMMARY:
The purpose of this study is to evaluate

1. the additional therapeutic benefit of Curodont Repair for the treatment early occlusal carious lesions on permanent teeth in children compared fluoride varnish alone
2. the tooth gel Curodont Protect when using it after Curodont Repair instead of fluoride varnish

DETAILED DESCRIPTION:
Objectives: The purpose of this study is to evaluate

1. the additional therapeutic benefit of Curodont Repair for the treatment early occlusal carious lesions on permanent teeth in children compared fluoride varnish alone
2. the tooth gel Curodont Protect when using it after Curodont Repair instead of fluoride varnish

Methods: 90 patients with early occlusal lesions (ICDAS-II:2-3) on permanent molars and pre-molars will be allocated in this randomized, controlled, single blinded study to one of the two test groups (Test1: Curodont™ Repair+Fluoride Varnish; Test2: Curodont Repair+Curodont Protect) or control (Fluoride Varnish) group.

Lesions will be assessed at baseline and recalls after 3, 6 and 12 months regarding caries activity (Nyvad), clinical status (ICDAS-II) and with Diagnodent®. Visual Analog Scale (VAS) in addition to the Global Impression of Change Questionnaire will also be used for the evaluation of the outcome.

ELIGIBILITY:
Inclusion Criteria:

* Early occlusal carious lesion which does not require an invasive treatment (ICDAS-II scores: 2 and 3)
* Size and form of the lesion: the lesion must both be fully visible and assessable and accessible
* Willing and able to attend the on-study visits and to observe good oral hygiene throughout the study
* Written informed consent before participation in the study

Exclusion Criteria:

* Evidence of tooth Erosion
* Fluoride varnish application < 3 months prior to study treatment
* History of head and neck illnesses (e.g. head/neck cancer)
* Any pathology or concomitant medication affecting salivary flow or dry mouth
* Any metabolic disorders affecting bone turnover
* Concurrent participation in another clinical trial

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Mean of values measured by Diagnodent(TM) (fluorescence measurement device for carious lesions) for each study group | Day 180
  Diagnodent values for fissure caries:
  0-5: no demineralization, sound. 6-14: outer enamel demineralization. 15-20: inner enamel demineralization. 21-99: dentine demineralization.

SECONDARY OUTCOMES:
Mean of values measured by Diagnodent(TM) (fluorescence measurement device for carious lesions) for each study group | Day 90 and Day 360
  Diagnodent values for fissure caries:
  0-5: no demineralization, sound. 6-14: outer enamel demineralization. 15-20: inner enamel demineralization. 21-99: dentine demineralization.
Frequency of change in ICDAS-II (International caries detection and assessment system) codes for each study group | Day 90, Day 180, Day 360
  Code 0: Sound tooth surface, no evidence of caries after prolonged air drying (5 sec).
  Code 1: First visual change in enamel. Code 2: Distinct visual change in enamel. Code 3: Localized enamel breakdown due to caries with no visible dentine or underlying shadow.
  Code 4: Underlying dark shadow from dentine with or without enamel breakdown. Code 5: Distinct cavity with visible dentine. Code 6: Extensive distinct cavity with visible dentine (involving more than half of the dentine).
Frequency of change in caries lesion activity and severity assessed by Nyvad criteria for each study group | Day 90, Day 180, Day 360
  Score 0: Sound. Score 1: Active caries - intact surface. Score 2: Active caries - surface discontinuity. Score 3: Active caries - cavity. Score 4: Inactive caries - intact surface. Score 5: Inactive caries - surface discontinuity. Score 6: Inactive caries - cavity.
Mean of VAS values (Visual analogue scale) for each study group | Day 90, Day 180, Day 360
  Range: from -50 (strongly remineralizing) to +50 (stronlgy progressing)
Frequency of Evaluation Outcome of Global Impression of Change Questionnaire for each study group | Day 90, Day 180, Day 360
  Investigator Questionnaire: evaluation ranging from "very much worse" to "very much better"; 7-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Dafina Doberdoli, Dr., Principal Investigator — University Dentistry Clinical Center of Kosovo